CLINICAL TRIAL: NCT05384418
Title: Cardiac AMyloidosis Prevalence and Outcome in Aortic Stenosis Patients Undergoing Transcatheter Aortic Valve Implantation (CAMPOS-TAVI)
Brief Title: Cardiac Amyloidosis Prevalence and Outcome in Aortic Stenosis Patients Undergoing Transcatheter Aortic Valve Implantation
Acronym: CAMPOS-TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PO20143
Record Dates: First submitted 2020-11-20; First posted 2022-05-20 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Aortic Stenosis
Keywords: Cardiac amyloïdosis; aortic stenosis; transthyretine amyloïdosis; CA-TTR; transcatheter aortic valve implantation; TAVI; prevalence; outcome; survival
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients undergoing transcatheter aortic valve implantation (Experimental): patients undergoing transcatheter aortic valve implantation for aortic stenosis
  Interventions: Radiation: HDP-Tc99m bone scintigraphy

INTERVENTIONS:
Radiation: HDP-Tc99m bone scintigraphy — HDP-Tc99m bone scintigraphy

SUMMARY:
Aortic stenosis (AS) is the most frequent valvulopathy in the general population in France and more generally in developed countries, due to populations aging. Its standard treatment is historically surgical aortic valve replacement (SAVR). In the 2000s, the management of this valvulopathy was revolutionized by the development of the technique of per-cutaneous aortic valve replacement (TAVI). TAVI opens the possibility of curative treatment to patients at high operational risk not operable by conventional surgery, and for whom outcome was affected with high mortality under medical treatment alone.

Amyloidosis, a pathology with multiple etiologies, is a rare condition and its cardiac form (AC) even more (8 to 17 / 100,000 people / year). However, its prevalence is increasing. Some autopsies series have found prevalence up to 50% of cardiac amyloidosis with transthyretin (AC-TTR) after 60 years. In addition, recent data suggested that AC-TTR prevalence is higher in the population of patients with heart disease: 13% in heart failure with preserved ejection fraction and up to 16% in patients with AS. The outcome of patients with AC-TTR remains unknown after TAVI. Thus, the diagnosis of AC-TTR in patients undergoing TAVI represents an important issue. Indeed, a treatment stabilizing the process of accumulation of transthyretin deposits, effective on the survival of these patients, is now available. In addition, a non-invasive screening strategy for AC-TTR, alternative to biopsy, is now validated.

DETAILED DESCRIPTION:
The aim of the study is to describe prevalence of cardiac amyloidosis with transthyretin in patients undergoing transcatheter aortic valve implantation.

ELIGIBILITY:
inclusion criteria :

* patients over 60 years old
* Patients admitted in Reims university cardiology department for per-cutaneous aortic valve replacement due to severe aortic stenosis
* Patients enrolled in the national healthcare insurance program
* Patients consenting to participate to the study

exclusion criteria :

- AL amyloïdosis patients

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2022-09-16 (Actual); Study Completion 2022-09-16 (Actual)

PRIMARY OUTCOMES:
transthyretine cardiac amyloïdosis | Hour 3
  Transthyretine cardiac amyloïdosis will be diagnosed using HDP-99mTc bone scintigraphy.
  The examination will consist of the injection of 10 MBq / kg of 99mTc-labeled biphosphonate, followed by a full-body scan 3 hours post-injection to produce a front thoracic static image and a tomographic image of the thorax.
  A positive HDP-Tc99m bone scintigraphy will be defined according to the Perugini classification corresponding to stages 2 and 3 (myocardial fixation of intensity equal to or greater than the bone structures).

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France